CLINICAL TRIAL: NCT05039866
Title: Long-Term Follow-up of Fabry Disease Subjects Who Were Treated With ST-920, an AAV2/6 Human Alpha Galactosidase A Gene Therapy
Brief Title: Long-Term Follow-up of Subjects Who Were Treated With ST-920
Status: Enrolling by invitation | Type: Observational
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ST-920-LT01
Record Dates: First submitted 2021-08-20; First posted 2021-09-10 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Fabry Disease; Fabry Disease, Cardiac Variant
Keywords: Fabry Disease; Gene Therapy; ST-920; Rare; Genetic; DNA; Sangamo; Long Term
MeSH Terms: conditions — Fabry Disease; Fabry Disease, Cardiac Variant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects who received ST-920: Subjects who received ST-920 in a separate parent trial
  Interventions: Biological: ST-920

INTERVENTIONS:
Biological: ST-920 — No study drug is administered in this study. Subjects who received ST-920 in a separate parent trial will be evaluated in this trial for long-term safety.

SUMMARY:
Long-term follow-up of subjects who received ST-920 in a previous trial (ST-920-201) and completed at least 52 weeks post-infusion follow-up in their primary protocol. Enrolled subjects will be followed for a total of up to 5 years following ST-920 infusion.

DETAILED DESCRIPTION:
Non-interventional, multi-center, long-term follow-up (LTFU) study of subjects dosed with ST-920 in the clinical study ST-920-201. All subjects dosed in the study who completed at least 52 weeks post-infusion follow-up in their primary protocol will be offered to participate. Subjects who enroll will be monitored for a total of up to 5 years following ST-920 infusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received ST-920 therapy in a separate parent trial
* Subjects who have consented to participate in this LTFU study.

Exclusion Criteria:

-This study has no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who have received ST-920 in separate parent trial and who have consented to participate in this Long Term Follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2039-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate long-term safety of ST-920 | 4 years
  To evaluate long-term safety of ST-920 by assessment of incidence and severity of adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sangamo Therapeutics, Inc.
Locations (13):
- United States (8):
  - University of California, Irvine, Irvine, California
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mt. Sinai Hospital, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Lysosomal & Rare Disorders Research & Treatment Center (LDRTC), Fairfax, Virginia
- The Royal Melbourne Hospital, Parkville, Victoria, Australia
- M.A.G.I.C. Clinic Ltd., Calgary, Alberta, Canada
- University Hospital of Würzburg, Würzburg, Germany
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - Royal Free Hospital, London